CLINICAL TRIAL: NCT03317353
Title: Reducing Rate of Falls in Older People With the Improvement of Balance by Means of Vestibular Rehabilitation: Preliminary Study
Brief Title: Reducing Rate of Falls in Older People by Means of Vestibular Rehabilitation: Preliminary Study
Acronym: ReFOVeRe
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Clinico Universitario de Santiago (Other)
Collaborators: Instituto de Salud Carlos III (Other Government); European Regional Development Fund (Other)
Responsible Party: Principal Investigator, Andrés Soto-Varela, Professor and Attending Physician, Hospital Clinico Universitario de Santiago
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: PI11/01328
Record Dates: First submitted 2017-10-18; First posted 2017-10-23 (Actual); Last update posted 2017-10-24 (Actual); Status verified 2017-10

CONDITIONS: Dizziness Chronic; Fall; Elderly
Keywords: Vestibular Rehabilitation; Falls in elderly; Computerized Dynamic Posturography; Optokinetic stimuli

STUDY DESIGN:
Intervention Model Description: Experimental study, single-center, open, randomized (balanced blocks of patients) in four branches in parallel, in 139 elderly patients (over 65 years) with high risk of falls; follow-up period: twelve months.
Who Masked: Investigator, Outcomes Assessor
Masking Description: Double (Investigator, Outcomes Assessor)
  After the first screening visit, the patients who grant their consent will be included in the study and randomised to one of the following study arms. Randomisation will be performed by C.H.U de Santiago Clinical Epidemiology and Biostatistics Unit. Once the informed consent form is signed, the care provider will contact the unit, which will give him the code of the arm to which the patient is assigned. A n= 20 block balanced randomisation sequence will be used. The investigator will analyse results and evolution, being blind type and duration of vestibular rehabilitation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Vestibular rehabil.: CDP (Experimental): Group A. The Smart Equitest program was used with a protocol of 10 exercises per session, which were customized depending on each patient´s deficit. The exercises involve visual biofeedback together with sensitive, real-time monitoring of movement. In some exercises, patients must maintain their center of gravity (COG) over the base of support, while in others the COG must be moved to a series of targets. In addition, the support surface and/or visual surround may also move in response to the patient´s own movement. The exercise difficulty was progressively increased throughout the rehabilitation sessions. The duration of each session was approximately 15 minutes. The distribution of sessions was one per day and five per week (2 weeks).
  Interventions: Device: Vestibular rehabil.: CDP
- Vestibular rehabil.: optokinetic stimuli (Experimental): Group B. Patient has to stand in a dark room, wiht optokinetic stimuli around him/her. Ten sessions (one per day, five per week, two weeks), with progressive increase of stimulus speed (from 30º/sec the first day to 100º/sec the last), duration of session (from 5 minutes the first day to 15 minutes the last), stimulus complexity (horizontal stimuli in the first sessions, progressively adding vertical and rotating stimuli) and support surface difficulty (initially hard surface, last sessions on foam).
  Interventions: Device: Vestibular rehabil.: optokinetic stimuli
- Vestibular rehabil.: home exercises (Experimental): Group C. The patient is given a list of exercises (and explained how to do them) to stabilise eye position and improve postural control. They are to be performed twice a day for two weeks. Approximate duration of each session: 15 minutes. The exercises must be supervised by a family member to verify adherence to the programme.
  Interventions: Other: Vestibular rehabil.: home exercises
- Control group (No Intervention): Group D. No vestibular rehabilitation is developed.

INTERVENTIONS:
Device: Vestibular rehabil.: CDP — Vestibular rehabilitation, ten sessions
  Other Names: Computerized Dynamic Posturography
  Arms: Vestibular rehabil.: CDP
Device: Vestibular rehabil.: optokinetic stimuli — Vestibular rehabilitation, ten sessions
  Arms: Vestibular rehabil.: optokinetic stimuli
Other: Vestibular rehabil.: home exercises — Exercises performed twice a day for two weeks. Approximate duration of each session: 15 minutes
  Arms: Vestibular rehabil.: home exercises

SUMMARY:
The aim of this study is to evaluate the effectiveness of vestibular rehabilitation to improve the balance in older people and reduce the number of falls, comparing three arms with different vestibular rehabilitation strategies (dynamic posturography exercises, optokinetic stimuli and exercises at home) and a control group.

DETAILED DESCRIPTION:
Vestibular rehabilitation has been shown to be effective in compensating patients with residual instability as a result of vestibular system disorders or Parkinson's disease. It is also useful for treating lack of balance in the elderly (presbivertigo). However, there is no systematic, controlled and prospective analysis of whether vestibular rehabilitation is effective in reducing the number of falls in the elderly, or whether its effects in this age group are temporary or persist over time.

This study compare vestibular rehabilitation with three different strategies (dynamic posturography exercises, optokinetic stimuli and exercises at home) and a control group, in people over 65 years. Balance tests are performed before vestibular rehabilitation and three weeks, six months and one year after it. Number of falls are quantified one year after vestibular rehabilitation.

ELIGIBILITY:
Inclusion Criteria:

Persons with a high risk of falling shall meet at least one of the following requirements:

* Having fallen at least once in the last 12 months.
* Using more than 15 seconds or needing support in the TUG test (normal limit calculated in previous studies).
* Obtaining a mean CDP SOT balance score of < 68% (normal limit calculated in previous studies).
* Having fallen at least once in the CDP SOT.

Exclusion Criteria:

* Cognitive decline that prevents the patient from understanding the examinations and vestibular rehabilitation exercises.
* Organic conditions that prevent standing on two feet, necessary for assessment of balance and performance of vestibular rehabilitation exercises.
* Balance disorders caused by conditions other than age (neurologic, vestibular...).
* Reduced cultural level that prevents the patient from understanding the examinations and from granting informed consent.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 139 (Actual)
Dates: Start 2012-01-01 (Actual); Primary Completion 2014-12-17 (Actual); Study Completion 2015-12-17 (Actual)

PRIMARY OUTCOMES:
CDP average | 12 months
  Average score in the Sensory Organization Test of the Computerized Dynamic Posturography

SECONDARY OUTCOMES:
Falls | 12 months
  Number of falls after vestibular rehabilitation
Hospitalisations | 12 months
  Hospitalisations due to falls in previous 12 months
DHI score | 12 months
  Dizziness Handicap Inventory score; it assesses the disability perceived by the patient in relation to instability. Minimum: 0; maximum: 100.
Short FES-I score | 12 months
  A shortened version of the falls efficacy scale-international to assess fear of falling score. Minimum: 0; maximum: 21.
Timed-up-and-go time | 12 months
  Duration (in seconds) of modified Timed-up-and-go test
Timed-up-and-go steps | 12 months
  Steps to perform the modified Timed-up-and-go test

CONTACTS AND LOCATIONS:
Overall Officials: Andrés Soto-Varela, PhD, Principal Investigator — Hospital Clinico Universitario de Santiago

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Rossi-Izquierdo M, Santos-Perez S, Del-Rio-Valeiras M, Lirola-Delgado A, Faraldo-Garcia A, Vaamonde-Sanchez-Andrade I, Gayoso-Diz P, Soto-Varela A. Is there a relationship between objective and subjective assessment of balance in elderly patients with instability? Eur Arch Otorhinolaryngol. 2015 Sep;272(9):2201-6. doi: 10.1007/s00405-014-3122-3. Epub 2014 Jun 12. PMID 24916738
- [Result] Soto-Varela A, Faraldo-Garcia A, Rossi-Izquierdo M, Lirola-Delgado A, Vaamonde-Sanchez-Andrade I, del-Rio-Valeiras M, Gayoso-Diz P, Santos-Perez S. Can we predict the risk of falls in elderly patients with instability? Auris Nasus Larynx. 2015 Feb;42(1):8-14. doi: 10.1016/j.anl.2014.06.005. Epub 2014 Sep 4. PMID 25194853
- [Result] Soto-Varela A, Gayoso-Diz P, Rossi-Izquierdo M, Faraldo-Garcia A, Vaamonde-Sanchez-Andrade I, del-Rio-Valeiras M, Lirola-Delgado A, Santos-Perez S. Reduction of falls in older people by improving balance with vestibular rehabilitation (ReFOVeRe study): design and methods. Aging Clin Exp Res. 2015 Dec;27(6):841-8. doi: 10.1007/s40520-015-0362-z. Epub 2015 Apr 25. PMID 25911608
- [Result] Rossi-Izquierdo M, Santos-Perez S, Faraldo-Garcia A, Vaamonde-Sanchez-Andrade I, Gayoso-Diz P, Del-Rio-Valeiras M, Lirola-Delgado A, Soto-Varela A. Impact of obesity in elderly patients with postural instability. Aging Clin Exp Res. 2016 Jun;28(3):423-8. doi: 10.1007/s40520-015-0414-4. Epub 2015 Jul 18. PMID 26187012
- [Result] del-Rio-Valeiras M, Gayoso-Diz P, Santos-Perez S, Rossi-Izquierdo M, Faraldo-Garcia A, Vaamonde-Sanchez-Andrade I, Lirola-Delgado A, Soto-Varela A. Is there a relationship between short FES-I test scores and objective assessment of balance in the older people with age-induced instability? Arch Gerontol Geriatr. 2016 Jan-Feb;62:90-6. doi: 10.1016/j.archger.2015.09.005. Epub 2015 Sep 18. PMID 26412554
- [Result] Soto-Varela A, Rossi-Izquierdo M, Faraldo-Garcia A, Vaamonde-Sanchez-Andrade I, Gayoso-Diz P, Del-Rio-Valeiras M, Lirola-Delgado A, Santos-Perez S. Balance Disorders in the Elderly: Does Instability Increase Over Time? Ann Otol Rhinol Laryngol. 2016 Jul;125(7):550-8. doi: 10.1177/0003489416629979. Epub 2016 Feb 4. PMID 26848036
- [Result] Faraldo-Garcia A, Santos-Perez S, Rossi-Izquierdo M, Lirola-Delgado A, Vaamonde-Sanchez-Andrade I, Del-Rio-Valeiras M, Soto-Varela A. Posturographic limits of stability can predict the increased risk of falls in elderly patients with instability? Acta Otolaryngol. 2016 Nov;136(11):1125-1129. doi: 10.1080/00016489.2016.1201591. Epub 2016 Jul 4. PMID 27376710
- [Result] Soto-Varela A, Faraldo-Garcia A, Del-Rio-Valeiras M, Rossi-Izquierdo M, Vaamonde-Sanchez-Andrade I, Gayoso-Diz P, Lirola-Delgado A, Santos-Perez S. Adherence of older people with instability in vestibular rehabilitation programmes: prediction criteria. J Laryngol Otol. 2017 Mar;131(3):232-238. doi: 10.1017/S0022215116009932. Epub 2017 Jan 16. PMID 28088930
- [Result] Rossi-Izquierdo M, Gayoso-Diz P, Santos-Perez S, Del-Rio-Valeiras M, Faraldo-Garcia A, Vaamonde-Sanchez-Andrade I, Lirola-Delgado A, Soto-Varela A. Short-term effectiveness of vestibular rehabilitation in elderly patients with postural instability: a randomized clinical trial. Eur Arch Otorhinolaryngol. 2017 Jun;274(6):2395-2403. doi: 10.1007/s00405-017-4472-4. Epub 2017 Mar 1. PMID 28251319